CLINICAL TRIAL: NCT03925012
Title: BOUNCE to Health: A Healthy Lifestyle Program
Acronym: BOUNCE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Houston (Other)
Collaborators: United Health Foundation (Unknown)
Responsible Party: Principal Investigator, Norma Olvera, Principal Investigator, University of Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 16447-01
Record Dates: First submitted 2019-04-08; First posted 2019-04-23 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Childhood Obesity; Obesity; Physical Activity; Health Knowledge, Attitudes, Practice; Health Behavior
MeSH Terms: conditions — Pediatric Obesity; Obesity; Motor Activity; Behavior; Health Behavior | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Child participants will attend the healthy lifestyle summer program for 4 weeks, five days per week. The summer intervention will include daily one-hour nutrition education, one-hour behavioral counseling, and 3 one-hour exercise sessions. These physical activities include flexibility, games, traditional fitness, and dancing. Counseling and school psychology students, registered dietitian/nutrition educators, and fitness specialists will lead the respective sessions. Parental guardians will participate in a two-hour weekly parental sessions that involve: 1)nutrition education with cooking demonstrations of healthy recipes; 2)behavioral counseling to learn effective parenting strategies on how to support their child's healthy nutrition and exercise habits and goals; and 3)exercise sessions where parents will engage in different physical activities and will receive fitness tips on how to promote an active lifestyle for the entire family.
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Intervention

SUMMARY:
The primary purpose of the BOUNCE study is to assess the effectiveness of a four-week family-based healthy lifestyle summer program in reducing adiposity indicators in Hispanic and African American girls and boys (ages 9-14 years old).

DETAILED DESCRIPTION:
The secondary aims of this study are to examine post-intervention changes in eating patterns, body image disturbances, unhealthy weight control practices, and fitness levels.

The investigators hypothesize that at the post-BOUNCE summer intervention, children will exhibit significant decreases in adiposity indicators (percent body fat and waist circumference), sweetened drinks and fried foods consumption, and an increase in physical fitness (aerobic capacity and minutes of moderated-vigorous physical activity) when compared to their baseline values after controlling for demographic, acculturation characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Both parental guardians (mother and father) and target child must be of Hispanic or African American descent
* Child must be between the ages of 9-14 years
* Child must be overweight/obese as defined by a body mass index percentile for age- gender specific between the 85th-100th percentile
* Child must have no physical disability or medical conditions that interfere with their participation in an exercise program
* Children must have no extensive diet restrictions that would hinder their participation in the BOUNCE nutrition component (e.g., unable to eat solid foods)
* All children will be required to submit evidence of a medical examination conducted by a health professional
* Parental guardians and child must be available to participate for the duration of the BOUNCE summer

Exclusion Criteria:

* Child and parental guardians are not Hispanic or African American
* Child is not between the ages of 9-14 years
* Child is underweight or normal weight (BMI < 85 percentile) or are morbidly obese (BMI > 100 percentile)
* Child or mother are pregnant or physically unable to participate
* Child has extensive diet restrictions that would hinder their participation in the BOUNCE nutrition component (e.g., unable to eat solid foods)
* Child does not have submitted evidence of a medical examination conducted by a health professional

Note: We will encourage both maternal and paternal guardians to participate in the measurements and interventions. However, if the paternal guardian refuses to participate or there is no father figure present in the family, maternal guardian-child pairs will be still eligible to participate in this study. If the children are of mixed race, but identify themselves as Hispanic or African American and at least one of their parents is either Hispanic or African American, they will be still eligible to participate.

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 720 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in Percent Body Fat | pre & post intervention at Week 4
  percent body fat obtained from a foot-to-foot bio-electrical impedance assessment
Anthropometric Change in Abdominal Fat | pre & post intervention at Week 4
  assessed through waist circumference (WC) measurements following guidelines from National Health and Nutrition Examination
Anthropometric Change in Hip Circumference | pre & post intervention at Week 4
  hip circumference (HC) measurements following guidelines from National Health and Nutrition Examination (for parents only)

SECONDARY OUTCOMES:
Physical Activity | pre & post intervention at Week 4
  Motion analyzer measures the percentage of youth who meet 60 minutes of daily moderate-to-vigorous physical activity per week
Sweetened Drinks | pre & post intervention at Week 4
  self-report measure
Fried Food Consumption | pre & post intervention at Week 4
  self-report measure

CONTACTS AND LOCATIONS:
Overall Officials: Norma Olvera, PhD, Principal Investigator — University of Houston
Locations (1):
- University of Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No